CLINICAL TRIAL: NCT06956443
Title: The Predictive Value of Quantified Indocyanine Green Fluorescent Angiography for Skin Necrosis in Mastectomy With Immediate Reconstruction
Brief Title: Prediction of ICG for Skin Necrosis in Mastectomy With Immediate Reconstruction
Status: Not yet recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Martini Hospital Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: nr. 2025-015
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancers; Mastectomy and Breast Reconstruction; Skin Necrosis
Keywords: ICG; mastectomy; breast cancer; breast reconstruction; skin necrosis
MeSH Terms: conditions — Breast Neoplasms; Necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICG group: All patients (those undergoing mastectomy with immediate breast reconstruction) belong to the same cohort.

SUMMARY:
Background Breast cancer represents 30 percent of newly diagnosed malignancies in female patients and is the leading cause of death in middle-aged women. Surgical treatment of breast cancer is performed with breast-conserving surgery or mastectomy. An increasing proportion of breast cancer patients undergo breast reconstruction after mastectomy. Reconstruction can be performed using various techniques that may involve the use of autologous tissues, implants, or a combination of both. However, mastectomy followed by immediate reconstruction can be associated with complications, including skin and fat necrosis, which occurs in 20% of cases.

When assessing tissue perfusion during immediate reconstruction, the surgeon relies on subjective observations, including skin color, capillary refill, and the occurrence of bleeding. One possible technique to assist the surgeon in assessing tissue perfusion is near-infrared (NIR) fluorescence imaging with Indocyanine Green (ICG). ICG can visualize tissue perfusion, because once in the bloodstream it is completely and permanently fixed to plasma proteins and circulates only in the intravascular compartment. ICG was approved for clinical use of tissue perfusion as early as 1956, such as in intestinal anastomoses, for the perfusion of free flaps or parathyroid glands.

ICG can also help predict postoperative skin necrosis in breast reconstruction after mastectomy. In patients undergoing (reconstructive) breast surgery, the intraoperative use of ICG NIR fluorescence imaging has been shown to help surgeons assess skin viability, thereby reducing the occurrence of skin necrosis in several studies. This reduction in necrosis can be explained by the intraoperative removal of tissue with reduced fluorescence intensity, observed with ICG NIR fluorescence imaging. However, there is no consensus on which ICG-NIR perfusion parameter is most accurate for assessing tissue perfusion. Further research is needed to determine cut-off values for adequate tissue perfusion. This study focuses on quantifying perfusion parameters and determining the diagnostic accuracy of ICG-NIR in patients undergoing mastectomy with immediate reconstruction.

What is the purpose of the study/research question? The purpose of this study is to determine the predictive value of quantified ICG fluorescence angiography for the occurrence of skin necrosis in patients undergoing mastectomy with immediate reconstruction with associated cut-off values.

Study design/procedure and intervention:

This will be a prospective cohort study of patients undergoing mastectomy with immediate reconstruction using ICG-NIR (the use of ICG during these operations is not an additional procedure).

This study will include patients who have undergone surgery with ICG (mastectomy with immediate reconstruction). We will use the videos of the ICG angiography for quantitative analysis of the data. This data will be correlated with the postoperative outcome (occurrence of skin/fat necrosis).

All patients will be asked in advance for permission to use their data. This will be processed pseudo-anonymously.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Patients undergoing mastectomy with immediate reconstruction using ICG-NIR
3. Patients are mentally competent
4. Written informed consent

Exclusion Criteria:

1. Patients with known allergy to ICG or iodinated contrast media
2. Pregnant or lactating women
3. Patients with dialysis-dependent renal failure and renal transplantation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing mastectomy with immediate reconstruction using ICG-NIR (as standard care) will be included if they meet the inclusion criteria. The treating surgeon will screen the patients and ask for their consent to use their data.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between occurrence of postoperative skin necrosis and quantified perfusion parameters | From enrollment to the end of analysis at 1 year and a half
  The occurrence of postoperative skin necrosis, defined as clinically evident necrosis of the mastectomy skin flap or subcutaneous fat, within the postoperative period.
  This will be correlated with quantified perfusion parameters obtained from intraoperative ICG-NIR fluorescence angiography, with the aim of determining the predictive value of these parameters.

SECONDARY OUTCOMES:
Diagnostic accuracy | From enrollment to the end of analysis at 1 year and a half
  Diagnostic accuracy of ICG-NIR fluorescence angiography in predicting postoperative skin necrosis, assessed by:
  Sensitivity
  Specificity
  Positive and negative predictive values
  Area under the receiver operating characteristic (ROC) curve (AUC)
Optimal cut-off values | From enrollment to the end of analysis at 1 year and a half
  Determination of optimal cut-off values for key ICG-NIR perfusion parameters (e.g., maximum fluorescence intensity, slope, time-to-peak, perfusion index), using ROC analysis, to differentiate between adequately and inadequately perfused tissue. The optimal cut-off values for perfusion parameters will be identified using Youden's index.